CLINICAL TRIAL: NCT01778452
Title: Profile Study of Genomics Endometrial Expression After Gonadotropin-releasing Hormone Agonist Administration and GnRH in Endometrial Priming.
Brief Title: Endometrial Genomic Profile in Endometrial Priming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VLC18012013
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Genomic Human Endometrial Expression Profile
Keywords: Endometrial priming, genomic expression. Natural cycle. Antagonist GnRH.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Natural cycle (Active Comparator): Natural cycle endometrial biopsy, lh+7
  Interventions: Procedure: endometrial biopsy
- Antagonist cycle + endometrial priming. (Experimental): Antagonist cycle + endometrial priming for egg donation program. endometrial biopsy, p4+5
  Interventions: Procedure: endometrial biopsy
- Agonist cycle + endometrial priming. (Experimental): Agonist cycle + endometrial priming for egg donation program endometrial biopsy, p4+5
  Interventions: Procedure: endometrial biopsy

INTERVENTIONS:
Procedure: endometrial biopsy — endometrial biopsy

SUMMARY:
The aim of this study is to analyse genomics profile expression in endometrium under different endometrial priming for recipients.

DETAILED DESCRIPTION:
We analyze the genomic profile of egg donors in different endometrial priming protocols, compared with natural cycle, including the conventional single long acting GnRH agonist injection in the mid luteal phase of the previous cycle of the endometrial priming and the single daily antagonist injection (Cetrorelix 0.25 mg) administered in the early follicular phase followed by endometrial priming. Endometrial biopsy will be taken in luteinizing hormone

* 7 or with P4 +5 in cases with endometrial priming with oestrogens therapy.

ELIGIBILITY:
Inclusion Criteria:

* 6 egg healthy volunteer egg donors.
* Volunteers.
* 18-35 years old
* Healthy.
* BMI <28.

Exclusion Criteria:

* - BMI > 28
* Smokers-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
genetic endometrial human profile expression | Oocyte donors will be followed up for four to six months
  implantation related genes profile expression

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Vidal, MDphD, Principal Investigator — IVI Valencia
Locations (1):
- Ivi Valencia, Valencia, Valencia, Spain